CLINICAL TRIAL: NCT01182168
Title: Phase I Trial of Gemcitabine and Split-Dose Cisplatin Plus Everolimus (RAD001) in Patients With Advanced Solid Tumor Malignancies
Brief Title: Gemcitabine and Split-Dose Cisplatin Plus Everolimus (RAD001) in Patients With Advanced Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-106
Record Dates: First submitted 2010-08-11; First posted 2010-08-16 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Bladder Cancer; Renal Pelvis Cancer; Ureter Cancer
Keywords: CISPLATIN; GEMCITABINE; RAD001 (EVEROLIMUS); 10-106
MeSH Terms: conditions — Urinary Bladder Neoplasms; Ureteral Neoplasms | interventions — Gemcitabine; Everolimus

ARMS (1):
- gemcitabine and cisplatin plus Everolimus (Experimental): This is a single-institution phase I study of gemcitabine and split-dose cisplatin plus escalating doses of continuous Everolimus (RAD001) in patients with advanced urothelial cancer.
  Interventions: Drug: gemcitabine and split-dose cisplatin plus escalating doses of continuous Everolimus (RAD001)

INTERVENTIONS:
Drug: gemcitabine and split-dose cisplatin plus escalating doses of continuous Everolimus (RAD001) — Patients will receive gemcitabine IV and cisplatin IV on days 1 and 8. Everolimus orally will be administered continuously (one cycle = 21 days). Everolimus will be escalated at the following dose levels: 5mg every-other-day, 5mg daily, and 10mg daily. Patients will receive a total of 6 cycles of gemcitabine and cisplatin in combination with Everolimus unless disease progression or unacceptable toxicity occurs.

SUMMARY:
The purpose of this study is to test the safety of gemcitabine and cisplatin plus Everolimus (also called RAD001) at different dose levels. We want to find out what effects, good and/or bad, this treatment has on you and your cancer.

Gemcitabine and cisplatin are standard chemotherapy drugs that are commonly used to treat advanced urothelial cancer. Everolimus is a pill that works by shutting down some of the pathways in cancer cells that make tumors grow. Laboratory studies have shown that Everolimus appears to improve the activity of cisplatin against cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have advanced urothelial cancer histologically confirmed by MSKCC pathology review.
* Patients may not have received prior systemic chemotherapy for metastatic disease.
* Patients may have received prior neoadjuvant or adjuvant systemic chemotherapy provided it was completed ≥ 1 year prior to the diagnosis of metastatic disease.

Age ≥ 18 years.

* Karnofsky Performance Status ≥ 70.
* Expected survival of at least 3 months.
* Resolution of all acute toxic effects of prior chemotherapy, radiotherapy, or surgical procedure to NCI CTCAE grade ≤ 1.
* Adequate bone marrow function as shown by:
* ANC ≥ 1.5x 109/L
* Platelets ≥ 100 x 109/L
* Hb >9 g/dL

Adequate liver function as shown by:

* Serum bilirubin ≤ 1.5 x ULN
* INR ≤ 1.5 (or < 3 on anticoagulants)
* ALT and AST ≤ 2.5x ULN (≤ 5x ULN in patients with liver metastases)

Adequate renal function as shown by:

* Serum creatinine ≤ 2.0 mg/dL OR

Calculated creatinine clearance ≥ 50 mL/min/1.73 m2 using the Jelliffe equation:

Calculated creatinine clearance = 98 - 0.8 [age(yrs) - 20] x (0.9 if female) Serum creatinine (mg/dL)

* Fasting serum cholesterol ≤ 300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: If a patient's lipid values exceed either one of these criteria upon screening, the patient can only become eligible after successful initiation of appropriate lipid-lowering medication. After lipid-lowering therapy, patients must meet the same criteria - i.e. a fasting serum cholesterol ≤ 300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN - to be eligible for study treatment.
* Testing for hepatitis B viral load and serological markers (HBV-DNA, HBsAg, HBsAb, and HBcAb) for the following patients:
* All patients who currently live in (or have lived in) Asia, Africa, Central and South America, Eastern Europe, Spain, Portugal, or Greece
* Patients with any of the following risk factors:
* Known or suspected past hepatitis B infection
* Blood transfusion(s) prior to 1990
* Current or prior IV drug users
* Current or prior dialysis
* Household contact with hepatitis B infected person(s)
* Current or prior high-risk sexual activity
* Body piercing or tattoos
* Mother known to have hepatitis B
* History suggestive of hepatitis B infection, e.g dark urine, jaundice, or right upper quadrant pain
* Additional patients at the discretion of the investigator
* Testing for hepatitis C infection (using quantitative RNA-PCR) for patients with any of the following risk factors:
* Known or suspected past hepatitis C infection (including patients with past interferon "curative" treatment)
* Blood transfusion(s) prior to 1990
* Current or prior IV drug users
* Household contact of hepatitis C infected person(s)
* Current or prior high-risk sexual activity
* Body piercing or tattoos
* Additional patients at the discretion of the investigator

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, tyrosine kinase inhibitors, etc.).
* Patients who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia), or patients who may require major surgery during the course of the study.
* Prior treatment with any investigational drug within the preceding 4 weeks.
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent, except corticosteroids with a daily dosage equivalent to prednisone ≤ 20 mg. Patients receiving these corticosteroids must have been on a stable dosage regimen for a minimum of 4 weeks prior to the first treatment with Everolimus. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period.
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
* Evidence of another active cancer, except for non-melanoma skin carcinoma, in-situ carcinoma of the cervix curatively treated, and adenocarcinoma of the prostate that has been surgically treated with a post-treatment PSA that is non-detectable.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as: symptomatic congestive heart failure of New York Heart Association Class III or IV.
* Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease.
* Severely impaired lung function as evidenced by:
* TLC <50% predicted OR
* FVC <50% predicted OR
* DLCO <40% predicted
* Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN.
* Active (acute or chronic) or uncontrolled severe infections.
* Liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis.
* A known history of HIV seropositivity.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of Everolimus (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Patients with an active, bleeding diathesis.
* Female patients who are pregnant or breast-feeding. Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to administration of Everolimus.
* Adults of reproductive potential who are not using effective birth control methods. Men and women of childbearing potential must be willing to use effective barrier method contraception during the trial and for at least 6 months thereafter. Patients are encouraged to continue barrier method contraception for two years or longer after treatment. Hormonal contraceptives are not acceptable as a sole method of contraception.
* Patients who have received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus).
* Patients with a known hypersensitivity to Everolimus (RAD001) or other rapamycins (sirolimus, temsirolimus) or to its excipients.
* Patients with a history of noncompliance to medical regimens.
* Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
To establish the dose-limiting toxicity (DLT) | 2 years
  of Everolimus in combination with gemcitabine and split-dose cisplatin in patients with advanced urothelial cancer.

SECONDARY OUTCOMES:
To establish the maximum tolerated dose (MTD) | 2 years
  of Everolimus in combination with gemcitabine and split-dose cisplatin in patients with advanced urothelial cancer.
To evaluate the response rate | 2 years
  of gemcitabine and split-dose cisplatin plus Everolimus in patients with advanced urothelial cancer and measurable disease as determined by RECIST.
To evaluate the time to disease progression | 2 years
  of gemcitabine and split-dose cisplatin plus Everolimus in patients with advanced urothelial cancer and measurable disease as determined by RECIST.
To assess activated mTOR pathway markers | 2 years
  in pre-treatment and post-treatment specimens, when available.
To evaluate overall survival | 2 years
  in patients with advanced urothelial cancer treated with gemcitabine and split-dose cisplatin plus Everolimus.
To assess activated PTEN status | 2 years
  in pre-treatment and post-treatment specimens, when available.
To assess activated Akt activation | 2 years
  in pre-treatment and post-treatment specimens, when available.
to evaluate markers of DNA repair | 2 years
  specifically BRCA1 and ERCC1 in pre-treatment and post-treatment specimens, when available.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Bajorin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm